CLINICAL TRIAL: NCT04497012
Title: Enteral Iron Supplementation and Intestinal Health in Preterm Infants
Brief Title: Iron Supplementation and Intestinal Health
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of South Florida (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Thao (Tina) Ho, Neonatologist, University of South Florida
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Pro00041470
Record Dates: First submitted 2020-07-20; First posted 2020-08-04 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-01

CONDITIONS: Anemia of Prematurity; Very Low Birth Weight Infant
Keywords: intestinal dysbiosis
MeSH Terms: conditions — Anemia | interventions — Iron-Dextran Complex

STUDY DESIGN:
Intervention Model Description: Randomize subjects to low and high dose iron supplementations
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The participants, care givers, medical teams, investigator, and outcome assessors are blinded from the iron treatment dose for the duration of the study. Only research pharmacists and members of the Data and Safety Monitor Board are unblinded during the study period.
  In an event when the medical team urgently needs to know the iron dose the participant is receiving for proper clinical management of the subject, the principal investigator or a designee will be notified by cell phone. Their contact information are located in the medical workrooms and the unit pharmacy. The principal investigator or the designee will immediately call the research pharmacy phone to request an emergency unblinding of that particular participant. The principal investigator will inform IRB and the sponsor of the unblinding event within 24 hours.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Low Iron Sulfate Supplementation (Active Comparator): Participants will be given 2 mg/kg/day total of elemental iron once a day when they are consuming 150-160 ml/kg/day of enteral feeds and are at least 14 days old. The total iron doses will be provided by fortification of feeds and liquid iron sulfate and will be weight adjusted once a week. The participants will receive the study iron dose until 36 week corrected gestational age or discharge, whichever comes first.
  Interventions: Drug: 2mg/kg/day Iron Sulfate
- High Iron Sulfate Supplementation (Active Comparator): Participants will be given 6 mg/kg/day total of elemental iron once a day when they are consuming 150-160 ml/kg/day of enteral feeds and are at least 14 days old. The total iron doses will be provided by fortification of feeds and liquid iron sulfate and will be weight adjusted once a week. The participants will receive the study iron dose until 36 week corrected gestational age or discharge, whichever comes first.
  Interventions: Drug: 6 mg/kg/day Iron Sulfate

INTERVENTIONS:
Drug: 2mg/kg/day Iron Sulfate — Iron Sulfate will be given in liquid form via nasal or oral gastric tube with feeds.
  Other Names: Low dose iron supplementation
  Arms: Low Iron Sulfate Supplementation
Drug: 6 mg/kg/day Iron Sulfate — Iron Sulfate will be given in liquid form via nasal or oral gastric tube with feeds.
  Other Names: High dose iron supplementation
  Arms: High Iron Sulfate Supplementation

SUMMARY:
This is a randomized double-blinded study of enteral iron supplementation in Very Low Birth Weight infants. The subjects will be randomized into low dose (2 mg/kg/day) and high dose (6 mg/kg/day) of daily iron supplementation. The primary outcomes are intestinal health including microbiome, inflammation, and barrier function.

DETAILED DESCRIPTION:
Infants and mothers will be recruited at a single academic level III NICU at Tampa General Hospital, Tampa, FL. Inclusion criteria infants: <1500 g at birth, expected to live beyond 2 weeks, not yet started on oral iron supplementation (OIS), and parental consent. Exclusion criteria infants: congenital intestinal defects, history of intestinal infection or perforation before OIS. Infants who require epogen for religious reason to prevent them from getting blood transfusions will be excluded from the study.

Intervention: Participants will be randomized to either 6 mg/kg/day or 2 mg/kg/day total of elemental iron once a day when they are consuming 150-160 ml/kg/day of enteral feeds and are at least 14 days old. The total iron doses will be provided by fortification of feeds and liquid iron sulfate and will be weight adjusted once a week. The participants will receive the study OIS doses until 36 week corrected gestational age or discharge, whichever comes first.

Sample collection and testing:

1. Stool and urine collection: We will collect weekly stool and urine samples non-invasively starting at enrollment until study completion. Samples will be collected from soiled diapers.
2. Blood tests: We will collect C-reactive protein (CRP) and ferritin level at 4 weeks after birth at the same time as other routine labs (complete blood count, reticulocyte count, and liver function test).
3. Monaural auditory brainstem response (ABR): for each ear will be performed at 36 weeks corrected gestational age or at discharge under the supervision of an audiologist who is blinded to the infants assigned iron doses and test results (stool microbiome, blood and urine tests).

Monitoring: iron supplementation dose will be increased by 2 mg/kg/day if ferritin level <100 mg/dL and the dose will be held if ferritin level >400 mg/dL. Ferritin level will be rechecked every 2 weeks until normalized. Hematocrit and reticulocyte count will be monitored by the medical team.

ELIGIBILITY:
Inclusion Criteria:

* <1500 g at birth, expected to live beyond 2 weeks, not yet started on oral iron supplementation (OIS), with mother at least 18 years of age, and parental consent.

Exclusion Criteria:

* congenital intestinal defects, history of intestinal infection or perforation before OIS. Infants who require epogen for religious reason to prevent them from getting blood transfusions will be excluded from the study.

Ages: 1 Day to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 183 (Estimated)
Dates: Start 2020-11-17 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in stool bacterial percentages from before to after iron supplementation | from baseline to 1 week and 2 weeks after iron supplementation started
  Comparing the changes in the median percentages of stool bacteria between the two groups. Change = post-iron (1 week, 2 weeks after iron and at discharge) - pre-iron
Change in fecal calprotectin from before to after iron supplementation | from baseline to 1 week and 2 weeks after iron supplementation started
  Comparing the mean fecal calprotectin levels, an inflammatory stool biomarker, between the two groups. Change = post-iron (1 week, 2 weeks after iron and at discharge) - pre-iron.
Change in urine Claudin-3 and I-FABP from before to after iron supplementation | from baseline to 1 week and 2 weeks after iron supplementation started
  Comparing the mean urine claudin-3 and I-FABP levels, biomarkers for intestinal barrier function, between the two groups. Change = post-iron (1 week, 2 weeks after iron and at discharge) - pre-iron

SECONDARY OUTCOMES:
Rate of auditory myelination | up to 36 weeks corrected gestational age
  Comparing the mean auditory latency levels between the two groups at 36 weeks corrected gestational age or at discharge.
Level of Iron storage | at 4 weeks after birth
  Comparing the mean Ferritin levels between the two groups at 4 weeks after birth

CONTACTS AND LOCATIONS:
Locations (1):
- Tampa General Hospital, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Strauss RG. Anaemia of prematurity: pathophysiology and treatment. Blood Rev. 2010 Nov;24(6):221-5. doi: 10.1016/j.blre.2010.08.001. PMID 20817366
- [Background] Mills RJ, Davies MW. Enteral iron supplementation in preterm and low birth weight infants. Cochrane Database Syst Rev. 2012 Mar 14;2012(3):CD005095. doi: 10.1002/14651858.CD005095.pub2. PMID 22419305
- [Background] Zimmermann MB, Chassard C, Rohner F, N'goran EK, Nindjin C, Dostal A, Utzinger J, Ghattas H, Lacroix C, Hurrell RF. The effects of iron fortification on the gut microbiota in African children: a randomized controlled trial in Cote d'Ivoire. Am J Clin Nutr. 2010 Dec;92(6):1406-15. doi: 10.3945/ajcn.110.004564. Epub 2010 Oct 20. PMID 20962160
- [Background] Jaeggi T, Kortman GA, Moretti D, Chassard C, Holding P, Dostal A, Boekhorst J, Timmerman HM, Swinkels DW, Tjalsma H, Njenga J, Mwangi A, Kvalsvig J, Lacroix C, Zimmermann MB. Iron fortification adversely affects the gut microbiome, increases pathogen abundance and induces intestinal inflammation in Kenyan infants. Gut. 2015 May;64(5):731-42. doi: 10.1136/gutjnl-2014-307720. Epub 2014 Aug 20. PMID 25143342
- [Background] Tang M, Frank DN, Hendricks AE, Ir D, Esamai F, Liechty E, Hambidge KM, Krebs NF. Iron in Micronutrient Powder Promotes an Unfavorable Gut Microbiota in Kenyan Infants. Nutrients. 2017 Jul 19;9(7):776. doi: 10.3390/nu9070776. PMID 28753958
- [Background] Krebs NF, Sherlock LG, Westcott J, Culbertson D, Hambidge KM, Feazel LM, Robertson CE, Frank DN. Effects of different complementary feeding regimens on iron status and enteric microbiota in breastfed infants. J Pediatr. 2013 Aug;163(2):416-23. doi: 10.1016/j.jpeds.2013.01.024. Epub 2013 Feb 26. PMID 23452586